CLINICAL TRIAL: NCT04738019
Title: A Multicenter, Prospective Observational Study to Evaluate the Incidence of Delayed-onset Nodules of YVOIRE Y-Solution 360, YVOIRE Y-Solution 540 or YVOIRE Y-Solution 720 Injected Into the Facial Skin Layer.
Status: Completed | Type: Observational
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-HAOS007
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy Condition
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Medical examination or treatment. — Medical examination or treatment when delayed on-set nodule or other side effects occur due to Y-Solution filler injection.

SUMMARY:
This is an observational study to evaluate the incidence of delayed-onset nodules of YVOIRE Y-Solution 360, YVOIRE Y-Solution 540 or YVOIRE Y-Solution 720 injected into the facial skin layer.

ELIGIBILITY:
Inclusion Criteria:

* Planned for YVOIRE Y-Solution 360 or 540 or 720 filler injection in facial area (except middle of the forehead, lips) for the volume enhancement or anti-wrinkle treatment.
* Male and female of 19 years or above age.
* Informed consent to participate in the study.
* Able to participate throughout the study period.

Exclusion Criteria:

* Prohibited in the Product Label.
* Have active or infectious skin disease in injection area.
* Autoimmune disease or HIV infected patient.
* Received immunosuppressive therapy within 2 weeks.
* Previously experienced Delayed-onset nodule after filler injection in facial area.
* Previously experienced Hypertrophic scar or Keloid.
* Have participated in an interventional clinical investigation within 30 days or plan to participate one during the study period.
* Ineligible for this clinical investigation as per Investigator's discretion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any healthy male and female whose filler injection on facial area is already planned for volume enhancement and anti-wrinkle treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Delayed-onset nodule. | 1 year.
  Incidence of delayed-onset nodule in the facial area Y-Solution 360 or 540 or 720 is injected.
Other adverse events. | 1 year.
  Other adverse events occur in the facial area Y-Solution 360 or 540 or 720 is injected.

CONTACTS AND LOCATIONS:
Locations (1):
- Dong Yeop Shin, Seoul, Gangseo-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Incidence rate of delayed-onset nodule or other side effects when YVOIRE Y-Solution 360 or 540 or 720 are used.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data is expected to be available during 2022.

REFERENCES:
- [Derived] Park SJ, Yoo KH. One-Year Safety Evaluation of New Hyaluronic Acid Fillers (YYS Series): A Prospective, Multicenter, Observational Study. Dermatol Surg. 2024 Aug 1;50(8):731-738. doi: 10.1097/DSS.0000000000004190. Epub 2024 May 2. PMID 38595129